CLINICAL TRIAL: NCT05111717
Title: The Effect of Desfluran Administered in General Anesthesia On Global Dna Methylation
Brief Title: The Effect of Desfluran On Global Dna Methylation
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Melike Korkmaz Toker, associate professor, Muğla Sıtkı Koçman University
Other Study IDs: MSKU 02/VII
Record Dates: First submitted 2021-10-17; First posted 2021-11-08 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: DNA Damage
Keywords: Desflurane,; DNA methylation; epigenetics; inhalation anesthetics
MeSH Terms: interventions — Desflurane

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral venous blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- group 1: Peripheral venous blood samples will collected at two time points as follows: before the premedication and the induction of anesthesia (T₁): 120 minutes after the beginning of anesthesia (T₂). DNA will be obtained from blood samples , and global DNA methylation analysis will be done.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Desflurane — Peripheral venous blood samplesof patients will collected at two time points as follows: before the premedication and the induction of anesthesia (T₁): 120 minutes after the beginning of anesthesia (T₂). Anesthesia maintenance will be provided with 40% O₂ and minimum alveolar concentration (MAC) in 60% air with 6% desflurane. DNA will be obtained from blood samples with the help of DNA isolation kit, and global DNA methylation analysis will performed by ELISA method.

SUMMARY:
The purpose of this study is to demonstrate the molecular effect of desflurane on DNA by measuring the global DNA methylation level in patients under going lumbar spinal stenosis surgery under general anesthesia.

DETAILED DESCRIPTION:
Forty patients scheduled for lumbar spinal surgery will include in the study. Peripheral venous blood samples will collect prior to the induction of anesthesia (T1) and after 120 minutes (T2). Anesthesia will maintaine with 40%-60% O2-air mixture and 6% desflurane. DNA will obtain from blood samples with the help of DNA isolation kit and global DNA methylation analysis will perform by ELISA method.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign an informed consent form
2. Elective lumbar spinal surgery that will take at least 120 minutes,
3. American Society of Anesthesiologists (ASA) physical status I and II
4. Be between the ages of 18 and 65

Exclusion Criteria:

1. Patients with ASA physical status III or IV disease
2. Smoking or alcohol consumption
3. Chronic systemic disease (diabetes mellitus,chronic pulmonary disorders, chronic kidney and liver disorders
4. recently received radiation, chemotherapy
5. malignancy
6. blood transfusion in operation
7. use of antioxidant supplements
8. have received general anesthesia in the last three months
9. Patients with known occupational exposures (operating room personnel, chemical plant workers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with physical status I and II of the American Society of Anesthesiologists (ASA), aged between 18-65 and scheduled for lumbar spinal surgery, which will take at least 120 minutes, will be included in the study
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Global DNA methylation change 5 minutes before and 120 minutes after anesthesia induction in peripheral blood mononuclear cells | 5 minutes before induction of anesthesia ,120 minutes after the beginning of anesthesia
  The global DNA methylation level will be measured 5 minutes before and 120 minutes after anesthesia induction.

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Sıtkı Kocman University Training and research Hospital, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
via mail

REFERENCES:
- [Background] Chowdhury B, Cho IH, Irudayaraj J. Technical advances in global DNA methylation analysis in human cancers. J Biol Eng. 2017 Mar 1;11:10. doi: 10.1186/s13036-017-0052-9. eCollection 2017. PMID 28261325
- [Background] Jaloszynski P, Kujawski M, Wasowicz M, Szulc R, Szyfter K. Genotoxicity of inhalation anesthetics halothane and isoflurane in human lymphocytes studied in vitro using the comet assay. Mutat Res. 1999 Feb 19;439(2):199-206. doi: 10.1016/s1383-5718(98)00195-8. PMID 10023059
- [Background] Bilban M, Jakopin CB, Ogrinc D. Cytogenetic tests performed on operating room personnel (the use of anaesthetic gases). Int Arch Occup Environ Health. 2005 Feb;78(1):60-4. doi: 10.1007/s00420-004-0579-1. Epub 2005 Feb 10. PMID 15703947